CLINICAL TRIAL: NCT00714350
Title: Evaluation of Information Displays A Paper & Pencil, Computer, Simulator, and ICU Based Study
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Noah Syroid, M.S., University of Utah
Other Study IDs: 23126; 2R44HL079783-02A1 (NIH)
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: Information Display; situational awareness; Create intuitive visualization

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Simulator Group - With Display: ICU nurses who viewed the new ICU display visualization
  Interventions: Behavioral: New ICU Display Visualization
- Simulator Group - Without Display: ICU nurses who did not view the new ICU display visualization, but instead viewed a traditional "spreadsheet" style presentation of ICU trends of data

INTERVENTIONS:
Behavioral: New ICU Display Visualization
  Groups: Simulator Group - With Display

SUMMARY:
Our objective is to develop intuitive, meaningful and ergonomically efficient informative displays specific to the user's domain. Specifically we aim to enhance and refine the display prototype of ABG information to include gas-exchange, acid-base balance, lung mechanics, ventilation, oxygenation, and metabolism information.

DETAILED DESCRIPTION:
To create an intuitive and meaningful visualization of Arterial Blood Gas (ABG) variables, it is necessary to address usability, ergonomics, domain specific, and expertise specific issues and concerns. Our objective is to develop intuitive, meaningful and ergonomically efficient informative displays specific to the user's domain. Specifically we aim to enhance and refine the display prototype of ABG information to include gas-exchange, acid-base balance, lung mechanics, ventilation, oxygenation, and metabolism information.

ELIGIBILITY:
Inclusion Criteria: ICU nurses Exclusion Criteria: All participants were screened and excluded from participation if they had previously participated in any of graphical display design and feedback sessions when developing the ICU display.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ICU nurses
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2007-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Nurses using the new ICU display will detect and communicate to an attending physician (confederate) more abnormal patient physiological states than when using the tabular (control) display. | At time of observation

CONTACTS AND LOCATIONS:
Overall Officials: Michael Behrens, Principal Investigator — University of Utah